CLINICAL TRIAL: NCT05010122
Title: A Phase I/II Study of ASTX727, Venetoclax, and Gilteritinib for Patients With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome With an Activating FLT3 Mutation
Brief Title: ASTX727, Venetoclax, and Gilteritinib for the Treatment of Newly Diagnosed, Relapsed or Refractory FLT3-Mutated Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0082; NCI-2021-06095 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0082 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-22; First posted 2021-08-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination; gilteritinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, cedazuridine, venetoclax, gilteritib) (Experimental): INDUCTION (CYCLE 1): Patients receive decitabine and cedazuridine PO QD on days 1-5, venetoclax PO QD on days 1-28, and gilteritinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity
  CONSOLIDATION (CYCLES 2-24): Patients receive decitabine and cedazuridine PO QD on days 1-5, gilteritinib PO QD on days 1-28, and venetoclax PO QD on days 1-14. Treatment repeats every 28 days.
  MAINTENANCE (CYCLES 24+): Patients receive gilteritinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Gilteritinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inqovi
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial studies the best dose of gilteritinib given together with ASTX727 and venetoclax and the effect of ASTX727, venetoclax, and gilteritinib in treating patients with FLT3-mutated acute myeloid leukemia that is newly diagnosed, has come back (relapsed) or does not respond to treatment (refractory) or high-risk myelodysplastic syndrome. Chemotherapy drugs, such as ASTX727, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Gilteritinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving ASTX727, venetoclax, and gilteritinib may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of the combination of decitabine and cedazuridine (ASTX727), venetoclax and gilteritinib in patients with relapsed/refractory FLT3- mutated acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS). (Phase I) II. To determine the complete response (CR)/incomplete hematologic recovery (CRi) rate of the regimen in patients with newly diagnosed or relapsed/refractory FLT3-mutated AML or high-risk MDS. (Phase II)

SECONDARY OBJECTIVES:

I. To assess other efficacy endpoints (CR rate, minimal residual disease negativity by flow cytometry, relapse-free survival, overall survival).

II. To assess proportion of patients proceeding to hematopoietic stem cell transplantation (HSCT).

III. To determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of baseline genomic alterations on response and survival of the combination regimen.

II. To determine the impact of baseline FLT3 allelic ratio on response and survival.

III. To evaluate clonal evolution from diagnosis to relapse using single-cell sequencing.

IV. To evaluate potential role of minimal residual disease (MRD) detection by sensitive polymerase chain reaction (PCR)/next generation sequencing (NGS) assays for FLT3 mutations.

V. To evaluate leukemia stem cell populations over the course of treatment with the combination regimen.

VI. To determine the impact of baseline apoptotic protein levels as assessed by mass cytometry (CyTOF) on response and resistance to the regimen.

OUTLINE: This is a phase I, dose-escalation study of gilteritinib followed by a phase II study.

INDUCTION (CYCLE 1): Patients receive decitabine and cedazuridine orally (PO) once daily (QD) on days 1-5, venetoclax PO QD on days 1-28, and gilteritinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity

CONSOLIDATION (CYCLES 2-24): Patients receive decitabine and cedazuridine PO QD on days 1-5, gilteritinib PO QD on days 1-28, and venetoclax PO QD on days 1-21. Treatment repeats every 28 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE (CYCLES 24+): Patients receive gilteritinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Phase I cohort: Adults >= 18 years with relapsed/refractory FLT3-mutated AML or myelodysplastic syndrome (MDS) that is intermediate-2 or high-risk by the International Prognostic Scoring System
  * Phase II cohort A: Adults >= 18 years with newly diagnosed FLT3-mutated AML. Patients should meet the following criteria:

    * Confirmed newly diagnosed AML with FLT3 mutation
    * Ineligible for induction therapy defined as

      * Either age >= 75
      * Or 18-74 with at least one comorbidity (congestive heart failure [CHF] requiring therapy or ejection fraction [EF] =< 50%, diffusion capacity of the lung for carbon monoxide [DLCO] =< 65% or forced expiratory volume in 1 second [FEV1] =< 65%, or Eastern Cooperative Oncology Group [ECOG] 2 or 3, or other significant co-morbidity precluding use of cytotoxic chemotherapy as approved by the principal investigator (PI)
  * Phase II cohort B: Adults >= 18 years with relapsed/refractory FLT3-mutated AML or MDS that is intermediate-2 or high-risk by the International Prognostic Scoring System who have received 1 prior therapy
  * For all cohorts, patients with either FLT3-ITD or FLT3 D835 mutations will be eligible
* Performance status =< 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the PI
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3 x ULN, unless due to the underlying leukemia approved by the PI
* Creatinine clearance >= 30 mL/min
* Ability to swallow
* Signed informed consent
* Hydroxyurea or one dose of cytarabine up to 1000 mg is allowed to reduce the white blood cell (WBC) to less than 25 x 10^9/L prior to initiation of study treatment

Exclusion Criteria:

* Prior therapies

  * Phase I cohort: No restriction based on prior therapies
  * Phase II cohort A: Patients with prior therapy for AML are not eligible. Prior therapy for antecedent hematologic disorder is allowed including prior hypomethylating agent (HMA) therapy for MDS. Prior hydroxyurea or cytarabine given for purposes of cytoreduction is also allowed. Prior all trans-retinoic acid given for presumed acute promyelocytic leukemia is also allowed
  * Phase II cohort B: Patients with >= 3 prior lines of therapy are not eligible. Stem cell transplantation, treatment given only for cytoreductive purposes (e.g. hydroxyurea), and growth factors do not count as lines of therapy for this purpose. Prior therapy with venetoclax and gilteritinib is allowed
* Patients suitable for and willing to receive intensive induction chemotherapy (for Phase II cohort A only)
* Congenital long QT syndrome or corrected QT (QTc) > 450 msec. Repeat electrocardiograms (EKGs) after correction of electrolytes or discontinuation of QT prolonging medications are allowed to meet entry criteria
* Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment)
* Active grade III-V cardiac failure as defined by the New York Heart Association Criteria
* Active central nervous system leukemia
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

  * Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
* Consumed strong inducer of CYP3A or p-glycoprotein within 3 days of study enrollment. Agents include but are not limited to: carbamazepine, phenytoin, rifampin, and St. John's wart
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids, hydroxyurea and/or cytarabine (given for cytoreduction) permitted. Use of hydroxyurea or one dose cytarabine to reduce WBC below 25 prior to initiation of study treatment is recommended
* Pregnant women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to use effective methods of contraception throughout the study period and for at least 6 months after the last dose of study drugs. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control throughout the study period and for at least 4 months after the last dose of study drugs. Lactating women (or those planning to breastfeed) should not breastfeed during treatment of gilteritinib and for at least 2 months after the last dose of gilteritinib
* Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I) | Up to 28 days
Overall response (OR) rate (Phase II) | Up to 2 cycles of treatment (1 cycle = 28 days)
  Will estimate the OR for the combination treatment (defined as the proportion of patients achieving complete response (CR) or incomplete hematologic recovery (CRi) within 2 cycles of treatment), along with the 95% credible interval.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Will also be estimated along with 95% credible interval.
To assess minimal residual disease negativity by flow cytometry | Up to 2 years
  Will also be estimated along with 95% credible interval.
Relapse-free survival | From the date of response to the date of documented relapses from CR or death from any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using the method of Kaplan and Meier.
Overall survival | From treatment start till death or last follow-up, assessed up to 2 years
  Will be estimated using the method of Kaplan and Meier.
Proportion of patients proceeding to hematopoietic stem cell transplantation | Up to 2 years
  Will also be estimated along with 95% credible interval.
Incidence of adverse events | Up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States